CLINICAL TRIAL: NCT01530217
Title: Assessing of Tooth Sensitivity Using Ibuprofen Before in Office-tooth Bleaching: a Randomized, Triple-blind Clinical Trial
Brief Title: Assessing of Tooth Sensitivity Using Ibuprofen Before in Office-tooth Bleaching
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidade Estadual de Ponta Grossa (Other)
Collaborators: Fundação Araucária (Other)
Responsible Party: Principal Investigator, Alessandra Reis, Doctor. Adjunctive Professors. School of Dentistry. State University of Ponta Grossa, Ponta Grossa, Paraná, Brazil., Universidade Estadual de Ponta Grossa
Allocation: Not Applicable | Model: Single Group | Masking: Triple | Purpose: Treatment
Other Study IDs: 17836/2010
Record Dates: First submitted 2011-12-13; First posted 2012-02-09 (Estimated); Last update posted 2012-02-09 (Estimated); Status verified 2012-02

CONDITIONS: Inflammation; Pulpitis
Keywords: Analgesics; Ibuprofen; Inflammation; Tooth Bleaching
MeSH Terms: conditions — Inflammation; Pulpitis | interventions — Ibuprofen

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: Ibuprofen. — Ibuprofen Group will be receive a dose of non-steroidal antiinflammatory drug ibuprofen 400 mg. All the participants will be watched to ensure that they took the drugs 1 hour prior to treatment. A second dose of ibuprofen (400 mg), will be administered a every 8 hours after the first dose during 48 hours.
  Other Names: Uniprofen / National Pharmaceutical Chemistry União S / A.

SUMMARY:
Ibuprofen has been recognized as anti-inflammatory and analgesic. The purpose of this study is to determine the effect of ibuprofen 400 mg on tooth sensitivity (TS) caused by in-office bleaching.

Methods: 30 health adults who received either placebo or ibuprofen. The drugs were administered 1 hour prior to the bleaching and will be prescribed 5 doses every 8 hours during 48 hours. For bleaching will be used 35% hydrogen peroxide gel. The tooth sensitivity will be recorded for up and lower arc on two scales: VAS (visual analogic scale) and 0-4. The shade evaluation will be performed before and 30 days after bleaching with visual shade guide and spectrophotometer.

DETAILED DESCRIPTION:
Background: Ibuprofen has been recognized as anti-inflammatory and analgesic. The purpose of this study was to determine the effect of ibuprofen 400 mg on tooth sensitivity (TS) caused by in-office bleaching.

Methods: A triple-blind, parallel design, randomized clinical trial will be conducted on 30 health adults who received either placebo or ibuprofen. The drugs will be administered 1 hour prior to the bleaching and a every eight hours during 48 hours. For bleaching used 35% hydrogen peroxide gel. The TS will be recorded for up and lower arc on two scales: VAS and 0-4. The shade evaluation will be performed before and 30 days after bleaching with visual shade guide and spectrophotometer. The % of patients that reported TS at least once during treatment and the TS intensity will be evaluated by Fisher's and Mann-Whitney tests, respectively. The color changes will be evaluated by repeated measures ANOVA.

ELIGIBILITY:
Inclusion Criteria:

* patients included in this clinical trial were:
* at least 18 years old.
* had good general and oral health.
* the participants should have eight caries-free maxillary and jaw anterior teeth and without restorations on the labial surfaces.
* the central incisors should be shade C2 or darker.

Exclusion Criteria:

* participants that had undergone tooth-whitening procedures.
* presenting anterior restorations.
* pregnant/lactating.
* with severe internal tooth discoloration (tetracycline stains, fluorosis, pulpless teeth).
* taking any kind of medicine, bruxism habits or any other pathology that could cause sensitivity (such as recession, dentine exposure).
* participants that reported some earlier or present health problems in stomach, heart, kidney and liver, or participants using any continuous drug with anti-inflammatory and antioxidant action were excluded from the study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2011-03; Primary Completion 2011-04 (Actual); Study Completion 2011-05 (Actual)

PRIMARY OUTCOMES:
Tooth sensitivity evaluation | Sensitivity during the treatment and until 48 hours after bleaching. The tooth sensitivity will be evaluated only this period because the literature appoint dates in this time.
  Patients will be distributed in two groups: Group 1 - Control Group will receive placebo. Group 2 - Ibuprofen will receive not selective anti-inflammatory (Ibuprofen 400 mg). All of the drugs will be administered one hour before the bleaching treatment. Evaluation of Dental Sensitivity Level: the effect of the product will be evaluated up to 1 Hour, 24 and 48 hours after the tooth bleaching, using a verbal scale of 5 points and a Visual Analogue Scale (VAS) will be used.

SECONDARY OUTCOMES:
Shade evaluation | Shade evaluation was recorded before and 30 days after the bleaching treatment.
  Shade evaluation was recorded using two methods: the subjective evaluation using a shade guide (Vita Lumin, Vita Zahnfabrik, Bad Säckingen, Germany) and an objective evaluation using the spectrophotometer (Easyshade, Vident, Brea, CA, USA).

CONTACTS AND LOCATIONS:
Overall Officials: Alessandra Reis, doctor, Principal Investigator — Universidade Estadual de Ponta Grossa